CLINICAL TRIAL: NCT05487300
Title: Effect of Levodopa on Cardiovascular Autonomic Function in Parkinson's Disease With and Without Orthostatic Hypotension: a Cross-over Study
Brief Title: Effect of Levodopa on Cardiovascular Autonomic Function in Parkinson's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Guillaume Lamotte, Assistant Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 00152581
Record Dates: First submitted 2022-07-29; First posted 2022-08-04 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease; Orthostatic Hypotension
MeSH Terms: conditions — Parkinson Disease; Hypotension, Orthostatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testing on-levodopa first, then off-levodopa (Other): Participants underwent autonomic testing one hour after taking their regular morning dose of levodopa (ON state). On a separate day, they then underwent autonomic testing after at least 12 hours from the last dose of levodopa (OFF state).
  Interventions: Drug: Autonomic testing on and off levodopa
- Testing off-levodopa, then on-levodopa (Other): Participants underwent autonomic testing after at least 12 hours from the last dose of levodopa (OFF state). On a separate day, they then underwent autonomic testing one hour after taking their regular morning dose of levodopa (ON state).
  Interventions: Drug: Autonomic testing on and off levodopa

INTERVENTIONS:
Drug: Autonomic testing on and off levodopa — Participants with Parkinson's disease with and without orthostatic hypotension will undergo standardized autonomic testing on two separate days "on levodopa" and "off levodopa".

SUMMARY:
Levodopa is a precursor of dopamine and is the treatment of choice to treat the motor symptoms of Parkinson's disease (PD); however, the effect of levodopa on cardiovascular autonomic function in PD is poorly understood. Orthostatic hypotension has been documented as a potential side effect of levodopa. As a result, clinicians may be reluctant to prescribe levodopa in patients with PD with neurogenic orthostatic hypotension (PD+OH), which leads to suboptimal management of motor symptoms. On the other hand, other studies failed to show any clear relationship between levodopa and orthostatic hypotension in patients with PD. Important limitations of prior studies include the lack of detailed investigation of baroreflex cardiovagal and sympathetic noradrenergic functions and the fact that the same patients were not tested on and off levodopa.

The investigators propose to investigate the effects of levodopa on cardiovascular autonomic function in patients with PD+OH and PD without neurogenic orthostatic hypotension (PD-OH) by performing standardized autonomic testing in the same patients on and off levodopa.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is characterized by the gradual onset of motor symptoms such as bradykinesia, rigidity, tremor, gait difficulties and postural instability, as well as non-motor symptoms such as cognitive impairment and autonomic dysfunction among others. Neurogenic orthostatic hypotension (nOH) is the main clinical manifestation of cardiovascular autonomic dysfunction. The arterial baroreflex allows for beat-to-beat regulation of the blood pressure and heart rate via differential modulation of its cardiovagal (parasympathetic) and noradrenergic (sympathetic) efferent limbs. Several mechanisms may contribute to nOH in PD including baroreflex-cardiovagal and baroreflex-sympathetic noradrenergic failure. The prevalence of nOH in PD increases with age and disease duration; however, several studies have documented that nOH may appear early in the course of PD and reported prevalence of nOH in PD ranges from 30% to 65%. The presence of nOH in PD is associated with poor outcomes related to cardiovascular events, increased morbidity and mortality, more rapid disease progression, cognitive impairment, and falls.

Levodopa is a precursor of dopamine and is the treatment of choice to treat the motor symptoms of PD; however, the effect of levodopa on cardiovascular autonomic function in PD is poorly understood. Orthostatic hypotension has been documented as a potential side effect of levodopa in different studies. As a result, clinicians may be reluctant to prescribe levodopa in patients with PD with nOH (PD+OH), which leads to suboptimal management of motor symptoms. On the other hand, several studies failed to show any clear relationship between levodopa and orthostatic hypotension in patients with PD. Important limitations of prior studies include the lack of detailed investigation of baroreflex cardiovagal and sympathetic noradrenergic functions and the fact that the same patients were not tested on and off levodopa.

The investigators propose to investigate the effects of levodopa on cardiovascular autonomic function in patients with PD+OH and PD without nOH (PD-OH) by performing standardized autonomic testing in the same patients on and off levodopa.

Clinical assessment: We will perform a medical history and physical examination before the testing procedures (baseline visit). The baseline visit will be performed on levodopa. The scales and assessments will include the Composite Autonomic Symptoms Score 31 (COMPASS 31), the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part I, II, III, and Hoehn and Yahr stage. The clinical assessment and scales are part of the standard of care in PD. Orthostatic vital signs will active standing will be also performed the two days of autonomic testing.

Participants will undergo a baseline visit. During the baseline visit, investigators will perform a medical history and physical examination and complete the following scales: Composite Autonomic Symptoms Score 31 (COMPASS 31), the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part I, II, III, and Hoehn and Yahr. Participants will undergo autonomic testing on two separate days. The first autonomic testing will occur within 4 weeks of the baseline visit. The two autonomic tests will occur within a 2-week timeframe. To avoid any confounding of treatment effects and period effects, the order of testing (on versus off levodopa) will be randomized so testing on the first day will be on-levodopa for half of the participants and off-levodopa for the other participants. Autonomic testing will include assessment of heart rate and blood pressures responses during the Valsalva maneuver and a 10-minute tilt table test.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of Parkinson's disease
* For the subgroup of participants with orthostatic hypotension (OH), OH will be defined by a sustained drop in systolic blood pressure > 20 mmHg and/or a drop in diastolic blood pressure > 10 mmHg within 3 minutes from supine to standing during tilt not attributable to medications. Autonomic testing and a ratio of orthostatic heart rate change/systolic blood pressure change < 0.5 bpm/mmHg will confirm the neurogenic etiology.

Exclusion Criteria:

* Any medication indicated for withdrawal that would result in undue risk to the participant if discontinued or that would confound heart rate and blood pressure measures
* Cognitive impairment that limits the ability to follow instructions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty individuals with PD (21 PD with orthostatic hypotension, 19 PD without orthostatic hypotension) were prospectively enrolled from August 1, 2022 to March 1, 2023. One subject did not complete visits 2 and 3 because of an unexpected surgery that was unrelated to the study and was excluded from the analysis. Another subject was excluded from the final analysis as a result of possible residual medication effects.
Period: Overall Study
Arm/Group | Testing On-levodopa First, Then Off-levodopa | Testing Off-levodopa, Then On-levodopa
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: One subject in the "Testing on-levodopa first, then off-levodopa" arm did not complete autonomic testing because of an unexpected surgery that was unrelated to the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Testing On-levodopa First, Then Off-levodopa | Testing Off-levodopa, Then On-levodopa | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 3
  >=65 years | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (8) | 73 (8) | 73 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 20 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39
Duration of disease [Number; unit: years] | 7.7 | 7.7 | 7.7

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure From Supine to Tilt at 3 Minutes
Description: Change in systolic blood pressure from supine to tilt at 3 minutes
Time Frame: from supine (baseline) to tilt at 3 minutes
Population: The results are presented ON vs OFF levodopa
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Testing ON Levodopa: Participants underwent autonomic testing one hour after taking their regular morning dose of levodopa (ON state).
- Testing Off Levodopa: Participants underwent autonomic testing after at least 12 hours from the last dose of levodopa (OFF state).
Arm/Group | Testing ON Levodopa | Testing Off Levodopa
Number analyzed (Participants) | 38 | 38
mmHg | -24.22 (17.69) | -20.32 (19.88)

2. Secondary Outcome: Baroreflex Cardiovagal Function
Description: Index of cardiovagal function: cardiovagal baroreflex sensitivity (BRS-V) [lower scores = worse outcome]. The BRS-V is the slope of the relationship between cardiac R-R interval and blood pressure in phase II of the Valsalva maneuver
Time Frame: Measure during Valsalva maneuver during autonomic testing (on levodopa and off levodopa)
Population: BRS-V - Results ON vs OFF levodopa
Measure: Mean (Standard Deviation); unit: ms/mmHg
Groups:
- Testing On-levodopa: Participants underwent autonomic testing one hour after taking their regular morning dose of levodopa (ON state)
- Testing Off-levodopa: Participants underwent autonomic testing after at least 12 hours from the last dose of levodopa (OFF state)
Arm/Group | Testing On-levodopa | Testing Off-levodopa
Number analyzed (Participants) | 38 | 38
ms/mmHg | 2.49 (2.39) | 2.02 (2.16)

3. Secondary Outcome: Baroreflex Adrenergic Sensitivity
Description: Baroreflex adrenergic sensitivity (BRS-A) in mmHg/s [lower scores = worse outcome]. The BRS-A was calculated as the systolic blood pressure decrement associated with phase 3 of the Valsalva maneuver divided by the blood pressure recovery time
Time Frame: BRS-A was calculated during the Valsalva maneuver (on and off levodopa)
Population: BRS-A - ON vs OFF levodopa
Measure: Mean (Standard Deviation); unit: mmHg/s
Arm/Group | Testing ON Levodopa | Testing Off Levodopa
Number analyzed (Participants) | 38 | 38
mmHg/s | 5.29 (6.51) | 6.88 (6.73)

ADVERSE EVENTS:
Time Frame: 1 day per each intervention through study completion, on average 3 weeks
Groups:
- Testing On-levodopa: Participants will undergo autonomic testing one hour after taking their regular morning dose of levodopa.
  Autonomic testing on and off levodopa: Participants with Parkinson's disease with and without orthostatic hypotension will undergo standardized autonomic testing on two separate days "on levodopa" and "off levodopa".
- Testing Off-levodopa: Participants will undergo autonomic testing at least twelve hours after taking their last dose of levodopa.
  Autonomic testing on and off levodopa: Participants with Parkinson's disease with and without orthostatic hypotension will undergo standardized autonomic testing on two separate days "on levodopa" and "off levodopa".
Arm/Group | Testing On-levodopa | Testing Off-levodopa
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT05487300/Prot_SAP_001.pdf